CLINICAL TRIAL: NCT02546544
Title: Phase II Trial of Linsitinib (Anti-IGF-1R/IR) in Patients With Relapsed and/or Refractory Ewing Sarcoma
Brief Title: Eurosarc Trial of Linsitinib in Advanced Ewing Sarcoma
Acronym: LINES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); European Commission (Other); Astellas Pharma Inc (Industry); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_038; 2012-000616-28 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2015-09-11 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2017-10

CONDITIONS: Relapsed Ewing Sarcoma; Refractory Ewing Sarcoma
Keywords: Linsitinib; anti-IGF-1R/IR; Ewing Sarcoma; dual IGF-1R/IR inhibition; Relapsed Ewing Sarcoma; Refractory Ewing Sarcoma; Metastatic Ewing Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Linsitinib (Other): Linsitinib is to be taken orally once a day on days 1-3, 8-10 and 15-17 on a 21 day cycle. The starting dose is 600 mg
  Interventions: Drug: Linsitinib

INTERVENTIONS:
Drug: Linsitinib
  Other Names: OSI-906; ASP7487

SUMMARY:
This is an international, multi-centre, single arm Bayesian designed phase 2 study to identify and determine the safety and activity of anti-IGF-1/IR inhibition in patients with relapsed and/or refractory ESFT. Approximately 40 patients will be recruited from 5-7 European centres. Each patient will be treated with single agent linsitinib, 600 mg orally once a day for days 1-3, 8-10 and 15-17 on a 21 day cycle until disease progression or undue toxicity.

DETAILED DESCRIPTION:
An important development in ES has been the identification of IGF-1R pathway dependency. The reasons for the remarkable single agent efficacy observed in a small subset of patients remains unknown, as is the relative lack of efficacy in the majority of patients. There may be heterogeneity in response due to partial signal pathway inhibition at the tumour level, inherent resistance in ES cells or the presence of alternative pathway activation through IR-A receptor signalling.

Here we aim to establish pharmacodynamic responses in ES tumours using functional imaging 18FDG-PET-CT and repeat post treatment biopsy for biomarker responses, toxicity and clinical outcome to the dual anti-IGF-1R/IR kinase blocking single agent linsitinib.

This is a single arm phase 2 study utilising adaptive Bayesian analysis. Approximately 40 patients will be recruited the national bone sarcoma centre in 5 EU countries over 18 months.

Eligible patients will take 4x 150 mg tablets once a day, days 1-3 of the week followed by 4 days off - repeated for 3 weeks = one treatment cycle. Patients can remain on treatment for as long as they gain clinical benefit.

The primary objectives are to determine the effect of linsitinib on the patient's tumours in terms of changes in biomarker and PET scans and to establish the safety of the trial drug (linsitinib) in Ewing sarcoma at the dose and treatment schedule being used in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed original (no new biopsy required) diagnosis of Ewing sarcoma, preferably with EWSR in situ hybridisation break apart probe.
* First, second or any relapse or refractory disease to conventional treatment
* Current disease state for which there either is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Has recovered from prior chemotherapy-related toxicity to ≤ grade 2
* Male or female, Age ≥ 18 and ≤70 years
* Life expectancy of at least 4 months
* WHO performance score of 0-2
* Must be able to take oral medication
* Is willing and able to comply with the protocol for the duration of the study, and scheduled visits and examinations, including biopsies and PET-CT scans
* Written (signed and dated) informed consent
* Tumour at biopsy accessible site; in the case of lung metastases, accessible with VATS procedure
* Tumour progression documented with imaging in the 6 months prior to study entry
* At least one measurable lesion on CT scan performed in past 14 days of minimum size 1 cm and 18FDG uptake positive
* Cardiac Ejection Fraction (Echocardiogram) ≥45%
* Fasting glucose ≤ 150 mg/dL (8.3 mmol/L) with no history of diabetes. Concurrent use of non-insulinotropic anti-hyperglycaemic therapy for diabetes is permitted if the dose has been stable for ≥ 4 weeks at the time of enrolment
* 16. Haematological and biochemical indices within the specified ranges as below:

  * Haemoglobin (Hb) ≥9 g/dL (Previous transfusion is allowed)
  * Absolute neutrophil count (ANC) ≥1.0 x 109/L without growth factor support
  * Platelet count > 80.x 109/L (Previous transfusion is allowed)
  * Direct Bilirubin <1.5 times the upper limit of normal (ULN)
  * Serum alanine aminotransferase (ALT) <2.5 x ULN for age and ≤ 5 x ULN if liver metastasis
  * Aspartate aminotransferase (AST) <2.5 x ULN for age
  * Alkaline phosphatase <2.5 x ULN for age
  * CPK <2.5 x ULN for age
  * Serum creatinine ≤1.5 x ULN for age
  * Potassium, magnesium and calcium within normal limits (supplementation and re-testing is permitted)

Exclusion Criteria:

* Females: Pregnant or breast-feeding, or of childbearing potential unless effective methods of contraception are used. Males: Unless effective methods of contraception are used.
* Significant active cardiac disease including: History (within last 6 months) of significant cardiovascular disease unless the disease is well-controlled. Significant cardiac disease includes second/third degree heart block; clinically significant ischemic heart disease; superior vena cava (SVC) syndrome; poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea).
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (≥ grade 3), left bundle branch block (LBBB), or asymptomatic sustained ventricular tachycardia are not allowed. Patients with atrial fibrillation controlled by medication are not excluded; uncontrolled high blood pressure (no greater than 2 SD above the mean for age for SBP and DBP), unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, or serious cardiac arrhythmias
* Mean QTcF interval ≥ 450 msec based on analysis of screening visit and pre-dose ECGs.
* 5. Use of drugs that have a known risk of causing Torsades de Pointes (TdP) within 14 days prior to registration
* Use of the potent CYP1A2 inhibitors ciprofloxacin and fluvoxamine within 7 days prior to registration. Linsitinib is primarily metabolized by CYP1A2 and inhibitors/inducers of CYP1A2 could alter the pharmacokinetics of linsitinib. Other less potent CYP1A2 inhibitors/inducers are not excluded
* Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results
* Any other active malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions
* History of cerebrovascular accident (CVA) within 6 months prior to entry that resulted in ongoing neurologic instability
* Patients with symptomatic brain metastases. Patients with previously diagnosed brain metastases are eligible if they have completed their CNS treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks, and are neurologically stable
* Major surgery within 4 weeks prior to study treatment
* Prior anti- IGF-1R treatment
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to enrolment
* Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Hassan, BMBCh FRCP, Principal Investigator — University of Oxford
Locations (5):
- Universitè Lyon 1 Claude Bernard, Lyon, France
- Pediatric Hematology and Oncology, University Hospital Münster, Münster, Germany
- Istituti Ortopedici Rizzoli, Bologna, Italy
- Department of Clinical Oncology, Leiden University Medical Center, Leiden, Postzone K1-P, Netherlands
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

REFERENCES:
- See also: Information about the trial on the Oncology Clinical Trials Office (OCTO) website. OCTO run the trial on behalf of the sponsor, the University of Oxford — http://www.octo-oxford.org.uk/alltrials/trials/LINES.html
- See also: ISRCTN registry — http://www.isrctn.com/ISRCTN94236001?q=cancer%20-radiotherapy&filters=recruitmentCountry:Netherlands&sort=&offset=21&totalResults=197&page=1&pageSize=100&searchType=basic-search

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from March 2014 until April 2016 at specialist cancer hospitals across Europe
Period: Overall Study
Arm/Group | Linsitinib
Started | 16
Received Allocated Intervention | 16
Completed | 0
Not Completed | 16
Not completed — Disease Progression | 14
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26.3 [24.1 to 28.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  Netherlands | 2
  United Kingdom | 8
  Italy | 4
  Germany | 2
WHO performance status [Count of Participants; unit: Participants] — The WHO performance status classification categorises patients as:
  0 able to carry out all normal activity without restriction
  1. restricted in strenuous activity but ambulatory and able to carry out light work
  2. ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours
  3. symptomatic and in a chair or in bed for greater than 50% of the day but not bedridden
  4. completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 5
    1 | 7
    2 | 4
Histology - Ewing Sarcoma [Count of Participants; unit: Participants] | 16
Primary site [Count of Participants; unit: Participants]
  Chest wall | 4
  Extra-osseous site | 2
  Lower extremity | 3
  Pelvis | 5
  Spine | 1
  Upper extremity | 1
Disease stage at screening - Metastatic [Count of Participants; unit: Participants] | 16
Sites of metastases [Number; unit: participants]
  Bone | 3
  Lung | 11
  Bone, Other | 8
Number of lines of previous treatment [Count of Participants; unit: Participants]
  Second line | 1
  Third line | 1
  > third line | 14
Time since most recent relapse/progression (days) [Median (Inter-Quartile Range); unit: days] | 18 [12 to 39]
Prior radiotherapy [Count of Participants; unit: Participants] | 13
Prior chemotherapy [Count of Participants; unit: Participants] | 16
Prior surgery [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Metabolic Response as Evaluated by PERCIST v1.0
Description: Metabolic response measured by PERCIST v1.0 using SULpeak. This methodology used SULpeak to measure change in glucose uptake in the tumour.
  Complete Metabolic Response - Complete resolution of 18F-FDG uptake within measurable target lesion so that it is less than mean liver activity and indistinguishable from surrounding background blood-pool levels.
  Partial Metabolic Response - Reduction of minimum of 30% in target measurable tumour 18F-FDG SULpeak. Absolute drop in SUL must be at least 0.8 SUL units, as well. No new lesions.
  Positive Metabolic Response - Participants having either "Complete Metabolic Response" or "Partial Metabolic Response".
  Stable Metabolic Disease - Not CMR, PMR or PMD. Progressive metabolic disease - Increase of more than 30% in 18F-FDG SUL peak. OR: Visible increase in extent of 18F-FDG tumour uptake (75% in TLG volume with no decline in SUL. OR: New 18F-FDG-avid lesions that are typical of cancer and not related to treatment effect or infection.
Time Frame: Pre- and Post- dose responses following 1 cycle (21 days) of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
Participants
  Positive metabolic response | 1
  Stable metabolic disease | 2
  Progressive metabolic disease | 4
  Not measurable at Baseline | 3
  Not assessable - liver | 4
  No repeat scan available | 2

2. Primary Outcome: Number of Participants With a Toxic Event
Description: A patient is defined as having a toxic event if they experienced at least one grade 3 adverse event (CTCAE v4.0 grade)
Time Frame: Following 6 cycles of treatment (up to 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
Participants
  Experienced a toxic event | 5
  Did not experienced a toxic event | 11

3. Secondary Outcome: Clinical Outcome (PFS, DSS)
Description: To determine the clinical outcome through assessment of
  * Progression free survival; where length of survival is defined in whole days as the time from entry into the study until Ewing sarcoma progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
  * Disease specific survival; where length of survival is defined in whole days as the time from entry into the study until death from Ewing sarcoma.
Time Frame: Duration of study (up to 18 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
months
  Disease specific survival | 7.1 [2.6 to NA] — Not enough participants achieved response to calculate upper 95% CI
  Progression free survival | 1.3 [0.7 to NA] — Not enough participants achieved response to calculate upper 95% CI

4. Secondary Outcome: Pharmacokinetics Assays of Following Linsitinib Treatment (Plasma Concentrations of Linsitinib)
Description: Plasma concentrations of linsitinib (ng/ml).
  Samples were taken 3 hours post-dose at Cycle 1 days 1,15,17, Cycle 2 day 3, Cycle 3 days 1 and 3, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1, and End of Treatment (this could occur at anytime during the 6 cycles).
Time Frame: Cycle 1 days 1,15,17, Cycle 2 day 3, Cycle 3 days 1 and 3, Cycle 4 day 1, Cycle 5 day 1, Cycle 6 day 1 and End of Treatment.0
Population: Data provided is as collected.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
ng/ml
  Screening: number analyzed (Participants) | 15
  Screening | 1 [1 to 1]
  Cycle 1 Day 1 | 4790 [286 to 7538]
  Cycle 1 Day 15: number analyzed (Participants) | 6
  Cycle 1 Day 15 | 2163 [1090 to 3206]
  Cycle 1 Day 17: number analyzed (Participants) | 11
  Cycle 1 Day 17 | 4977 [144 to 9628]
  Cycle 2 Day 3: number analyzed (Participants) | 2
  Cycle 2 Day 3 | 3409 [1534 to 5284]
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | 6791 [849 to 8478]
  Cycle 3 Day 3: number analyzed (Participants) | 5
  Cycle 3 Day 3 | 1964 [417 to 14080]
  Cycle 4 Day 1: number analyzed (Participants) | 1
  Cycle 4 Day 1 | 3591 [3591 to 3591]
  End of treatment visit: number analyzed (Participants) | 5
  End of treatment visit | 1 [1 to 1432]
  Cycle 5 Day 1: number analyzed (Participants) | 0
  Cycle 6 Day 1: number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With a Radiological Response as Evaluated by RECIST v1.1
Description: Radiological response measured using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)
  Per RECIST for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), >20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable disease (SD), Not CR, PR or PD.
Time Frame: Measured cycle 1 day 15, cycle 3 and cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
Participants
  Cycle 1: Stable disease | 7
  Cycle 1: Progressive disease | 7
  Cycle 1: No repeat scan available | 2
  Cycle 3: Stable disease | 2
  Cycle 3: Progressive disease | 4
  Cycle 3: No repeat scan available | 10
  Cycle 6: Stable disease | 0
  Cycle 6: Progressive disease | 0
  Cycle 6: No repeat scan available | 16

6. Secondary Outcome: Number of Participants With a Metabolic Response as Evaluated by EORTC 1.0
Description: as for outcome 1
Time Frame: Measured cycle 1 day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Linsitinib
Number analyzed (Participants) | 16
Participants
  Positive metabolic response | 2
  Stable metabolic disease | 5
  Progressive metabolic disease | 7
  No repeat scan available | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until 28 days post treatment.
Arm/Group | Linsitinib
All-Cause Mortality (participants affected / at risk) | 13/16
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linsitinib (N=16)
Diarrhoea (Gastrointestinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linsitinib (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 4
Pain (General disorders) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 6
Haemoglobin decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes